CLINICAL TRIAL: NCT05241756
Title: Femtosecond Laser-Assisted Cataract Surgery in Pediatric Patients, a Prospective Case Series
Brief Title: FLACS in Pediatric Patients Using FEMTO LDV-Z8
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziemer Ophthalmic Systems AG (Industry)
Responsible Party: Sponsor
Other Study IDs: CPFEM-0003-BE
Record Dates: First submitted 2022-01-12; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Cataract in Child
Keywords: FLACS; Femto-LDV Z8; Pediatric; Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- FLACS using FEMTO LDV-Z8
  Interventions: Device: FLACS using FEMTO LDV-Z8

INTERVENTIONS:
Device: FLACS using FEMTO LDV-Z8 — Performance of femtosecond laser-assisted capsulotomy in the anterior capsule.

SUMMARY:
This study is a single center prospective observational case series. The framework of this clinical investigation is post market clinical follow up of pediatric FLACS using the Femto LDV Z8. The intention is to investigate and supervise aspects particular to the pediatric use, and there is hence no alternative patient population.

Primary outcome Related adverse events at the time of surgery, ophthalmic adverse events at 1 week, 1 month, 6 months.

Secondary outcome Achieved vs aimed capsulotomy diameter

* Aimed diameter to be calculated using the Bochum formula
* Achieved diameter will be assessed using a ring caliper (Morcher 4.8 external diameter), (US patent MJ Tassignon)

During the recruitment period, the legal representatives of all patients (and when applicable the patients) at the study site who are eligible for pediatric cataract surgery and fulfilling the eligibility criteria will be informed about the study and offered participation. The aim is to include 12 participants during the recruitment period of 6 months. Inclusion criteria are on purpose chosen very broad, in order to collect data from all types of pediatric cataract surgeries.The majority of the participants will be very young children, who cannot be involved in the informed consent procedure. Participants will nevertheless receive the patient information in a way adapted to their age and mental maturity, from investigators or members of the investigating team who are experienced in working with children. The study procedure is cataract surgery performed with the FEMTO LDV Z8 femtosecond laser. In this clinical investigation the CE marked products (the Femto LDV™ femtosecond laser and the FEMTO LDV™ Surgical Laser Procedure Packs for Cataract Surgery) are used without deviations from the intended use and indication for use. Intraoperatively the achieved capsulotomy diameter will assessed using a ring caliper (Morcher 4.8 external diameter) and compared with the aimed diameter calculated using the Bochum formula. Patients will return for follow-up visits at 1 week, 1 month, 6 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 18 years at the time of surgery
2. In case of bilateral cataract, only one eye will be included in the study
3. Informed consent of the legal representative of the patient (and as applicable, the patient) documented per signature
4. Planned cataract surgery
5. Accurate baseline biometric measurements
6. Assessed medical status
7. Full pupil dilatation is achieved using Cyclopentolate eye drops

Exclusion Criteria:

1. Eyes with microphthalmia of < 9 mm diameter white to white
2. Hazy cornea
3. Pregnancy; girls of childbearing age will be tested for pregnancy with urinary analysis (hCG) at the time of inclusion.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients of Antwerp University Hospital assigned to undergo a cataract surgery.
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Number of intraoperative and postoperative adverse events | Up to 6 months
  Number of intraoperative and postoperative adverse events

SECONDARY OUTCOMES:
Aimed capsulotomy diameter | Done intraoperatively
  - Aimed diameter to be calculated using the Bochum formula
Achieved capsulotomy diameter | Done intraoperatively
  - Achieved diameter will be assessed using a ring caliper (Morcher 4.8 external diameter), (US patent MJ Tassignon)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-José Tassignon, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University and University Hospital Antwerp (UZA), Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No